CLINICAL TRIAL: NCT03163680
Title: Efficacy of Low Dose of Proton Pumb Inhabitor in Treatment Upper Gastrointestinal Bleeding
Brief Title: Efficacy of Low Dose of Proton Pump Inhibitor in Treatment Bleeding Ulcers
Status: Completed | Type: Observational
Sponsor: Damascus Hospital (Other)
Responsible Party: Principal Investigator, Marouf Alhalabi, MD, Damascus Hospital
Other Study IDs: G6-17
Record Dates: First submitted 2017-05-15; First posted 2017-05-23 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Gastroduodenal Ulcer; Marginal Ulcer; Peptic Ulcer Hemorrhage
Keywords: Gastroduodenal Ulcer; Marginal Ulcer; Peptic Ulcer Hemorrhage; Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer; Peptic Ulcer Hemorrhage | interventions — Omeprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low Dose PPI: patients with upper upper gastrointestinal bleeding were treated in low dose of proton Bump inhibitor meaning 40 mg twice daily
  Interventions: Drug: Omeprazole 40 MG

INTERVENTIONS:
Drug: Omeprazole 40 MG — Omperazole 40 mg twice daily

SUMMARY:
Determining the efficacy of low dose of PPI in management acute peptic ulcer bleeding

DETAILED DESCRIPTION:
Determining the efficacy of low dose meaning 40 mg of omeprazole twice in management acute peptic ulcer bleeding

ELIGIBILITY:
Criteria:

Inclusion Criteria:

High risk ulcers defined according to the Forrest classification With respect to high-risk stigmata, active bleeding was defined as a continuous blood spurting (Forrest IA) oozing (Forrest IB) from the ulcer base. A non-bleeding visible vessel at endoscopy was defined as a discrete protuberance at the ulcer base(Forrest IIA).

An adherent clot was one that was resistant to forceful irrigation or suction (Forrest IIB).

Exclusion Criteria:

ulcer was malignant non ulcerative bleeding such as angiodysplasia , a Mallory-Weiss tear

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the gastrointestinal department of damascus hospital
Sampling Method: Non-Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Morality | within 1 week
  Determination of mortality rate from ulcer bleeding

SECONDARY OUTCOMES:
Rebleeding | within 1 week
  Determination of the percentage of the return of bleeding represented by recurrent melena (black, tarry stool) or recurrent Hematemesis or coffee-ground emesis or recurrent hematochezia after begin treatment
need for surgery | within 1 week
  Determine the Surgery rate for treatment Bleeding ulcers within a week
Length of hospital stay | within 1 month
  Determining the length of stay in the hospital
Blood transfusions | within 1 week
  number of transfusion blood unites during admission

CONTACTS AND LOCATIONS:
Locations (1):
- Damascus Hospital, Damascus, Syria

IPD SHARING:
Plan to Share IPD: Undecided